CLINICAL TRIAL: NCT01459666
Title: A Prospective, Multi-Center, Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Efficacy of AbobotulinumtoxinA (BTX-A) in Improving Forehead Wounds After Mohs Micrographic Surgery and Reconstruction for Skin Cancer
Brief Title: Forehead Scars Following Mohs Micrographic Surgery and Reconstruction for Skin Cancer
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Investigator left institution for private practice
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Dr. Kevin Cooper, Principal Investigator, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CASE1Z12
Record Dates: First submitted 2011-10-18; First posted 2011-10-26 (Estimated); Results first posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-04

CONDITIONS: Scar
Keywords: Scar; Forehead; Skin Cancer; MOHS Surgery; Dermatology
MeSH Terms: conditions — Cicatrix; Skin Neoplasms | interventions — abobotulinumtoxinA; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dysport (abobotulinumtoxinA) (Experimental): Each patient will be able to receive up to 120 units of Dysport/placebo at the initial visit to treat the entire forehead area (the frontalis, procerus, and corrugator muscles) to insure cosmetic symmetry. Injections will be placed a minimum of 1.5cm above the orbital rim at the mid papillary line to minimize the risk of lid ptosis. The actual amount to be injected will be at the discretion of the Mohs surgeon based on his or her opinion of what amount is needed for sufficient wound paralysis and cosmetic symmetry.
  Interventions: Drug: Dysport (abobotulinumtoxinA)
- Placebo (Placebo Comparator)
  Interventions: Drug: Bacteriostatic 0.9% Sodium Chloride (vehicle)

INTERVENTIONS:
Drug: Dysport (abobotulinumtoxinA) — Intramuscular injection effects lasting up to 3 months
  Other Names: AbobotulinumtoxinA; Clostridium botulinum type toxin A toxin-haemagglutinin complex
  Arms: Dysport (abobotulinumtoxinA)
Drug: Bacteriostatic 0.9% Sodium Chloride (vehicle) — Intramuscular injection
  Arms: Placebo

SUMMARY:
This study will test if the use of DysportTM (abobotulinumtoxinA) improves wound healing and scarring after Mohs surgery. Research in the laboratory as well as previous studies in humans have shown improved wound healing and scarring with the use of a similar medication called Botox.

Dysport may improve wound healing and scarring by relaxing facial muscles and therefore minimizes the muscle tension and possibly the inflammation around the wound.

DETAILED DESCRIPTION:
Primary Objective:

-To evaluate the efficacy of using aboBTX-A to improve wound healing prior to Mohs micrographic surgery and reconstruction for skin cancer as measured by the Visual Analogue Scale (VAS) at 6 weeks post surgery.

Secondary Objectives:

* To evaluate efficacy of using aboBTX-A to improve wound healing prior to Mohs micrographic surgery and reconstruction for skin cancer as measured by the Patient and Observer Assessment Scale (POSAS) at week 1, 6, and 24.
* To evaluate the efficacy of using aboBTX-A to improve wound healing prior to Mohs micrographic surgery and reconstruction for skin cancer as measured by the Visual Analogue Scale (VAS) at week 1 and 24 post surgery.
* To evaluate patient satisfaction
* To evaluate safety (adverse events)

This is a 6 month, prospective, multicenter, double-blinded, randomized, placebo-controlled study. A total of 40 male or female healthy volunteers, 20 in each arm, will be enrolled. Up to 10 more patients can be enrolled to account for patient drop-out. Subjects will all undergo Mohs micrographic surgical removal of a skin cancer lesion on the forehead followed by reconstruction. Subjects will be randomized to receive either aboBTX-A injection or placebo injection in the frontalis, procerus, and corrugator muscles prior to reconstruction. Photographs, POSAS, and clinical assessments will be taken immediately after initial wound closure, at 1 week follow-up, at 6 weeks follow-up, and at 6 months follow-up. Adverse events will also be reviewed at each study visit. After the completion of the study, the photographs will be assessed (blinded as to the patient identifiers) using a 10 cm visual analog scale (VAS). The first few photographs will be evaluated by the surgeons together to calibrate the VAS and ensure inter-reliability.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be eligible for enrollment:

* Ability to understand the risks, benefits, and alternative to participation and give informed consent
* Have biopsy proven skin cancer on the medial forehead that is amenable to Mohs surgery. Medial forehead is defined as the area superiorly from the hairline, inferiorly at the eyebrow, and laterally to the tip of the lateral brow (see diagram).
* Undergoing elective reconstruction of biopsy proven skin cancer that is amenable to Mohs surgery with defect size measuring 1.0 cm or greater
* If female, not currently pregnant, no potential for pregnancy, or if of child-bearing age, must agree to use adequate contraception (e.g., hormonal or barrier method of birth control; abstinence) for 30 days after the last dose of study drug. A negative urine pregnancy test is required at study entry for female subjects of childbearing potential: a woman is considered to be of child bearing potential unless she has had a tubal ligation, total hysterectomy, bilateral oopherectomy, or is postmenopausal (without a menstrual period for at least one year)
* Agrees to not use disallowed concomitant medications (retinoids)

Exclusion Criteria:

The presence of any of the following will exclude a patient from study enrollment.

* Pregnant women, women who are breastfeeding, or women of child bearing age who are unwilling to use adequate contraception (described above) during the study period
* Current or past history of a neuromuscular disease (such as myasthenia gravis, amyotrophic lateral sclerosis, Eaton-Lambert syndrome)
* Currently taking aminoglycosides or other agents interfering with neuromuscular transmission (e.g., curare-like agents)
* History of radiation therapy or chemotherapy
* History of keloid or other hypertrophic scar formation
* Current or past history of scleroderma
* Has used botulinum toxin in the forehead area within one year.
* Has significant resting eyebrow ptosis
* Has used any topical retinoids to the forehead area within the past 4 weeks
* Undergo any scar revision procedure for the duration of the study including intralesional kenalog, laser treatment, and/or scar revision surgeries
* Any hypersensitivity to any component of abobotulinumtoxinA (i.e. cow milk protein) or any previous hypersensitivity to any botulinum toxin A or related product.
* Non-English speaking: These patients are excluded since translation of the informed consent into other languages is time-consuming and expensive as it requires a bona fide translator for the particular language of interest and this type of person may be difficult to locate.
* House staff and students, medical students on a clerkship, and employees related to study personnel or who work for any study personnel, and members of the study team are not eligible to participate in this study as a subject.
* The investigator feels that for any reason the subject is not eligible to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-09; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Mann, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (2):
- United States (2):
  - University Hospitals Cleveland Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - UH Cleveland Medical Center-Westlake, Westlake, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was terminated, only 9 participants were actually enrolled.
Period: Overall Study
Arm/Group | Dysport (abobotulinumtoxinA) | Placebo
Started | 5 | 4
Completed | 0 | 0
Not Completed | 5 | 4
Not completed — PI left institution | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dysport (abobotulinumtoxinA) | Placebo | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 3 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 4 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 4 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Scale (VAS)
Description: It consists of a 10 point scale to assess global scar assessment. Scar photographic images are assessed by independent physicians, and previous studies have shown very high intrarater consistency.
Time Frame: 6 weeks post surgery
Population: Not collected
Arm/Group | Dysport (abobotulinumtoxinA) | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Patient and Observer Assessment Scale (POSAS)
Description: The Patient and Observer Scar Assessment Scale (POSAS) consists of two numeric scales. One scale is completed by the patients, the other by the clinician. This scale is different than previous scales because it takes the patient's input into consideration. It has good internal consistency and interobserver reliability. The assessment will take place at Day 0, Week 1, Week 6, and Month 6.
Time Frame: at week 1, 6, and 24 post surgery
Population: Not collected
Arm/Group | Dysport (abobotulinumtoxinA) | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Visual Analogue Scale (VAS)
Description: Evaluate efficacy of using aboBTX-A to improve wound healing prior to Mohs micrographic surgery and reconstruction for skin cancer as measured by the Visual Analogue Scale (VAS)
Time Frame: at week 1 and 24 post surgery
Population: Not collected
Arm/Group | Dysport (abobotulinumtoxinA) | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 7 Months
Arm/Group | Dysport (abobotulinumtoxinA) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 0/5 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-10-23): https://cdn.clinicaltrials.gov/large-docs/66/NCT01459666/Prot_SAP_000.pdf